CLINICAL TRIAL: NCT02484820
Title: PREMAPESSAIRE: Prevention of Preterm Birth in Singletons Using Pessary After Resolutive Threatened Preterm Labor: a Prospective, Randomized Monocentric Clinical Trial
Brief Title: Prevention of Preterm Birth in Singletons Using Pessary After Resolutive Threatened Preterm Labor
Acronym: PREMAPESSAIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1508059; 2015-A00672-47 (Other: ANSM)
Record Dates: First submitted 2015-06-17; First posted 2015-06-30 (Estimated); Last update posted 2023-05-24 (Actual); Status verified 2023-02

CONDITIONS: Preterm Birth
Keywords: Preterm Birth; pessary; threatened preterm labor
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pessary (Experimental): Silicone pessary is associated with standard care Silicone pessary is used between 24 weeks of pregnancy and up to 6 weeks after the date of the term (maximum 6 months)
  Interventions: Device: Silicone pessary
- Control (No Intervention): Standard care only, No silicone pessary will be placed in the vagina.

INTERVENTIONS:
Device: Silicone pessary — Silicone pessary is used between 24 weeks of pregnancy and up to 6 weeks after the date of the term (maximum 6 months)
  Arms: Pessary

SUMMARY:
In France, threatened preterm labour concerns 6.5% of pregnancies and is associated with a premature birth in 25.4% of cases.

After 48 hours effective tocolysis, patients do not receive any further treatment while their risk of premature birth has risen from 6.5% to 25%.

A pessary is a silicone ring encircling the cervix. It was initially used as medical treatment of genital prolapse but studies were also conducted for pregnant women in 2 high-risk premature birth situations: cervical incompetence and twin pregnancies.

The multicenter PECEP trial conducted by Goya and al. in asymptomatic short cervix patients between 18 and 22 weeks of gestation showed a significant reduction of premature birth before 34 and 37 weeks of gestation. Thereby, the investigator assume that use of pessaries in patients presenting a resolutive threatened preterm labor will also be effective.

To evaluate this hypothesis, the investigator designed a randomized prospective single-center open clinical trial comparing pessary associated with standard care (1st group) versus standard care only (2nd group) in patients experiencing an episode of resolutive threatened preterm labor.

ELIGIBILITY:
Inclusion Criteria:

* Minimal age of 18 years
* Informed consent
* Confirmation of dating of pregnancy by first trimester echography.
* Episode of threatened preterm labour
* Singleton between 24 and 34 weeks of gestation
* Cervical length ≤20mm in cervimetry
* Pulmonary maturation completed
* ≤6 contractions by hour after 24 hours of tocolysis.

Exclusion Criteria:

* Major fetal abnormalities (requiring surgery or leading to infant death or severe handicap)
* Spontaneous rupture of membranes at the time of randomization
* Cervical cerclage in situ
* Uterus malformations
* Antecedent of conisation
* Active vaginal bleeding, placenta previa
* Intra-amniotic infection
* Hydramnios
* Maternal chronic pathology (hypertension, diabetes)
* Anomaly of breathing foetal rate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2022-10-08 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Number of spontaneous delivery | 37 weeks of gestation
  Comparison of the number of spontaneous delivery before 37 completed weeks of gestation for pregnant women after resolutive threatened preterm labour between 20 and 34 weeks of gestation between the 2 groups of the study.

SECONDARY OUTCOMES:
Number of spontaneous delivery | 34 weeks of gestation
  Comparison of the number of spontaneous delivery before 34 completed weeks of gestation for pregnant women after resolutive threatened preterm labour between 20 and 34 weeks of gestation between the 2 groups of the study.
Number of spontaneous delivery | 28 weeks of gestation
  Comparison of the number of spontaneous delivery before 28 completed weeks of gestation for pregnant women after resolutive threatened preterm labour between 20 and 34 weeks of gestation between the 2 groups of the study.
Number of admission for preterm labor | from date of randomization until the date of the delivery
  Comparison of the number of admission for preterm labor from date of randomization until the date of the delivery between the 2 groups.
Number of fetal-neonatal death | at delivery
  Number of fetal-neonatal death at delivery
Number of birth death | From date of delivery until 6 weeks after the date of term
  Number of birth death at delivery until 6 weeks after the date of term
Number of patients with neonatal morbidity | From date of delivery until 6 weeks after the date of term
  Number of patient with neonatal morbidity at delivery until 6 weeks after the date of term
Number of patients with increase of vaginal discharge | from date of randomization until the date of the delivery
  Comparison of the number of patients with increase of vaginal discharge from date of randomization until the date of the delivery between the 2 groups of the study.
Number of patients with spontaneous pessary ejection | from date of randomization until the date of the delivery
  Comparison of the number of patients with pessary ejection from date of randomization until the date of the delivery between the 2 groups of the study.
Number of patients with discomfort | from date of randomization until the date of the delivery
  Comparison of the number of patients with discomfort from date of randomization until the date of the delivery between the 2 groups of the study. The discomfort is measure by a standardized questionnaire.
number of day between resolutive threatened preterm labor and delivery | At delivery
  Comparison of number of day between the two groups of the study

CONTACTS AND LOCATIONS:
Overall Officials: Céline CHAULEUR, PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Chu Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No